CLINICAL TRIAL: NCT00528125
Title: Laser Acupuncture for Pain Prevention in Neonates Undergoing Heel Prick. A Prospective, Randomized, Double-blinded Clinical Trial
Brief Title: Laser Acupuncture for Pain Prevention in Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children Hospital Homburg (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SG-07-H-02
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2008-03

CONDITIONS: Pain
Keywords: pain prevention; neonatal pain; laser acupuncture; complementary and alternative medicine
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Active laser acupuncture
  Interventions: Procedure: active laser acupuncture
- B (Placebo Comparator): placebo laser acupuncture
  Interventions: Procedure: placebo laser acupuncture

INTERVENTIONS:
Procedure: active laser acupuncture — low level laser acupuncture, 830 nm, 30 mW, 0,3 J per acupoint, 2 points per neonate (Hegu and Shen Men). Overall 30 seconds of treatment
  Other Names: Modulas Handy 2/99, schwamedico, Ehringshausen, Germany
  Arms: A
Procedure: placebo laser acupuncture — placebo laser acupuncture at two acupoints (Hegu, Shen Men). Overall treatment time 30 seconds.
  Other Names: placebo laser, Modulas Handy 2/99, schwamedico, Ehringshausen, Germany
  Arms: B

SUMMARY:
Pain prevention and/or therapy in neonates is still a challenge. It is widely accepted that early pain experience can have a tremendous impact on the pain memory. We want to investigate if a simple, fast method, that is nearly devoid of side effects can lead to a significant alleviation of pain sensation in neonates. Acupuncture has been shown to be effective in various painful conditions. Trials on acupuncture in children are rare. Trials on acupuncture in neonates are lacking so far. Our hypothesis is that neonates in the active laser group experience less pain than those in the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with no obvious underlying disease (genetic (e.g. M. Down), metabolic)and not under pain medication

Exclusion Criteria:

* Older than 28 days

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
The Pain score Premature Infant Pain Profile (PIPP), according to video analysis | 5 minutes from the heel prick
  The Premature Infant Pain Profile (PIPP Score) is a reliable instrument to measure acute pain in neonates and it includes objective vital parameters and is not only a third-party observation. A total of seven indicators are measured: Three behavioural indicators (facial actions: eye squeeze, brow bulge and nasolabial furrow), two physiological indicators (heart rate and oxygen saturation), and two contextual indicators (gestational age and behavioral state). A scoring of 0, 1, 2 or 3 points is used for each of the seven indicators. All indicators are summed up to a total score. Depending on the gestational age, the possible total score ranges from 18 to 21.

SECONDARY OUTCOMES:
Cry Time | right after after heel prick up to 5 minutes
  in seconds (according to the Audio track of the video analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Gottschling, MD, Principal Investigator — University Children Hospital Homburg, Germany; Ludwig Gortner, MD, PhD, Study Director — University Children Hospital Homburg, Germany
Locations (1):
- University Children Hospital Homburg, Homburg, Saarland, Germany